CLINICAL TRIAL: NCT07192315
Title: Predicting Reactions and Effects of Drugs Immunotherapy and Complications Through Oncosafety (PREDICTO Clinical Study)
Acronym: PREDICTO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCAPHM25_0294; 2025-A01531-48 (Other: IDRCB)
Record Dates: First submitted 2025-07-21; First posted 2025-09-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor Malignancies; Solid Cancers
Keywords: immuno-induced adverse events; Immune checkpoint inhibitor; baseline predictive signature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood, Throat and skin swabs and Stool additional samples (Experimental): Blood, Throat and skin swabs and Stool additional samples are collected in parallel of treatment administration throughout visits 1 to 4.
  Interventions: Other: Bloodsampling; Other: Pharyngeal swab sampling; Other: Cuteanous swab sampling; Other: Stools sample collection

INTERVENTIONS:
Other: Bloodsampling — Blood will be sampled At Visit 1, 2, 3 and 4. For patients presenting immuno-induced adverse events (iRAEs), an additionnal visit V tox will be planned will a blood sampling.
Other: Pharyngeal swab sampling — Pharyngeal swab will be sampled at visit 4 for patients without immuno-induced adverse events (iRAEs) Pharyngeal swab will be sampled at visit Tox for patients presenting immuno-induced adverse events (iRAEs)
Other: Cuteanous swab sampling — Cuteanous swab will be sampled at visit 1, 2, 3 and 4 for patients without immuno-induced adverse events (iRAEs).
  Cuteanous swab will be sampled at visit 1, 2, 3 and tox for patients presenting immuno-induced adverse events (iRAEs).
Other: Stools sample collection — Stools sample will be collected at visit 1, 2, 3 and 4 for patients without immuno-induced adverse events (iRAEs).
  Stools sample will be collected at visit 1, 2, 3 and tox for patients presenting immuno-induced adverse events (iRAEs).

SUMMARY:
Immune Checkpoint Inhibitors (ICI) have revolutionized cancer therapy, providing unprecedented responses in a wide range of malignancies. However, they induced various immune-related adverse events (iRAE) that can be life-threatening. About 20% of patients treated with an ICI monotherapy, and up to 60% of patients treated with a combination of ICIs, experienced a severe iRAE. Most side effects are reversible if managed early, but can affect survival and quality of life, leading to treatment interruptions or hospitalization. Some of these irAEs, particularly those affecting hormonal functions, may be irreversible and persist even after treatment discontinuation.

The development of predictive biomarkers of such toxicities is an unmet medical need. The variety of mechanisms involved in iRAE, and the lack of effective animal models, could probably explain why the topic remains largely unexplored. To date, some biomarkers predictive of the occurrence of iRAE, irrespective of the type of organ affected, have been identified by state-of-the-art techniques on small cohorts prior to treatment initiation, but none is individually robust enough to be used in daily practice.

We hypothesize that a signature derived from the integrative analysis of various biological parameters (immunomonitoring, auto-immunity features, viral monitoring, microbiota monitoring, fragmentome analysis, pharmacokinetics, radiomics and genetics), available in routine hospital practice, could answer this question, and thus enable the development of specific prevention strategies

The objectives are :

Primary objective:

Identify a baseline predictive signature for severe iRAE, irrespective of the type of organ affected.

Secondary objectives:

* Identify a predictive signature for severe iRAE including baseline and T1 data, irrespective of the type of organ affected.
* Identify a baseline predictive signature for organ-specific severe iRAE.
* Identify a predictive signature for organ-specific severe iRAE including baseline and T1 data.
* Identify a baseline predictive signature for severe iRAE, irrespective of the type of organ affected, for patient receiving an anti-PD(L)1 in monotherapy.
* Identify a baseline predictive signature for severe iRAE, irrespective of the type of organ affected, for patient receiving an anti-PD(L)1 in combination.
* Identify a baseline predictive signature for severe iRAE, irrespective of the type of organ affected, for each specific immunotherapy received.
* Compare the predictive signatures between responders and non-responders according to RECIST 1.1 in order not to overlook the influence of clinical response on the variability observed.
* Describe the results obtained for each biological parameter between severe irAEs and non-severe irAEs patients.
* Describe patient-reported outcomes and quality of life parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Histologically or cytologically confirmed solid tumour malignancy
* Patients are included in the study before their first infusion of immunotherapy with anti-PD1, anti-PDL1, anti-CTLA4, anti-LAG3, alone or in combination, as part of standard care, in all validated solid oncology indications.
* Patient treated at AP-HM in one of the CEPCM-affiliated departments.
* Inclusions will be made such that at least 40% of included patients receive a combination of ICIs
* Ability to comply with study procedures and follow-up schedule
* The patient must have given free and informed consent and signed the consent form
* Patient must have at least one measurable lesion according to RECIST 1.1 criteria
* Patient who is a beneficiary or entitled beneficiary of a social security scheme

Exclusion Criteria:

* Patients previously treated with ICIs
* The patient's therapeutic plan includes targeted therapy, chemotherapy or any other systemic treatment in combination with ICI
* Patient has an active autoimmune disease or any other pathology requiring systemic corticosteroid therapy at more than 10 mg prednisone equivalent per day or any other immunosuppressive drug
* Patients with a history of organ transplantation, hematopathy or hematopoietic stem cell transplantation
* History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Patients of Adults without legal capacity
* Patients in Health and Social Establishments
* Persons in emergency situations
* Persons deprived of their liberty
* Absence or refusal of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Identification of a predictive baseline signature who maximize the rate of prediction of severe iRAE | From enrollment to the end of following after 12 months
  The primary endpoint is the identification of a predictive baseline signature who maximize the rate of prediction of severe iRAE among patients who had a severe iRAE (iRAE + patients) and minimize the rate of prediction of severe iRAE among patients who had not a severe iRAE (iRAE- patients), we choose a minimum of 70% of prediction in iRAE + population and a maximum of 15% of prediction in iRAE- population.

SECONDARY OUTCOMES:
Assesment of safety according to NCI-CTCAE v5.0 criteria | From enrollment to the end of following after 12 months
Identification of signatures for severe iRAEs | From enrollment to the end of following after 12 months
  Predictive performance of baseline + T1 signatures for severe iRAEs
Identification of signatures for organ-specific severe iRAEs | From enrollment to the end of following after 12 months
  Predictive performance of baseline signatures for organ-specific severe iRAEs using the same performance thresholds.
Identification of signatures for organ-specific severe iRAEs at baseline and T1 | From enrollment to the end of following after 12 months
  Predictive performance of baseline + T1 signatures for organ-specific severe iRAEs.
Identification of signatures for severe iRAEs in patients receiving anti-PD(L)1 monotherapy. | From enrollment to the end of following after 12 months
  Performance of baseline signatures for severe iRAEs in patients receiving anti-PD(L)1 monotherapy.
Identification of signatures in patients receiving combination immunotherapy | From enrollment to the end of following after 12 months
Identification of baseline signatures for each specific immunotherapy class. | From enrollment to the end of following after 12 months
Comparison of predictive signatures between responders and non-responders (RECIST 1.1). | From enrollment to the end of following after 12 months
Rate of biological parameter variation between severe and non-severe iRAE patients | From enrollment to the end of following after 12 months
Assessment of PRO-CTCAE | From enrollment to the end of following after 12 months
  NCI-PRO-CTCAE (Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events): which is a 81-item instruments designed to measure symptoms and side effects for patients through treatment for their cancer. Items are constructed on a 5-point Likert scale with the following response options: 1 "Not at all" / 2 "A little" / 3 "Quite a bit" / 4 "severe" / 5 "Extremely severe".
Evaluation of quality of life via EORTC QLQ-C30 questionnaire | From enrollement to the end of following after 12 months
  EORTC QLQ-C30 : European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire, which is a 30-item instrument designed to measure quality of life in all cancer patients. 28 items are constructed on a 4-point Likert scale with the following response options: 1 "Not at all" / 2 "A little" / 3 "Quite a bit" / 4 "A lot." The last two items are constructed on a 7-point response scale.
  These two items assess the patient's physical condition and overall quality of life, respectively, with response 1 corresponding to a "very poor" condition and response 7 to an "excellent".
Evaluation of quality of life via EQ-5D-5L questionnaire | From enrollement to end of the following after 12 months
  EQ-5D-5L, which is descriptive system EuroQol comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Scale frome 1 to 100, where 0 is the worst possible condition and 100 is the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided